CLINICAL TRIAL: NCT05956561
Title: Correlation Between Serum Vitamin D Level And Early Implant Failure
Brief Title: Correlation Between Vitamin D Serum Level and Early Implant Failure
Acronym: EDIF
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mona nady Abd El-Raouf, Mona Nady Abd El-Raouf, Ain Shams University
Other Study IDs: EDIF 863
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Endosseous Dental Implant Failure
Keywords: early implant failure; implant stability; vitamin D

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- only one group: all patients seeking delayed dental implant placement above 18 years and medical free, no previous augmentation or sinus lifting
  Interventions: Other: dental implants were placed for all cases while assessing vitamin D levels

INTERVENTIONS:
Other: dental implants were placed for all cases while assessing vitamin D levels — vitamin D assessment with measuring implant stability and clinical finding of early failure

SUMMARY:
The goal of this observational study is to investigate relation between serum vitamin D levels and early implant failure. in all patient seeking delayed dental implant placement at Faculty of Dentistry, Ain Shams University from September 2020 to April 2023, all the patients must fulfil the inclusion criteria including age above 18, no medical condition interference and compliance to study. The main question[s] it aims to answer are:

* is vitamin D deficiency caustic to early implant failure
* can implant stability indicate implant failure Participants will receive implants and prosthetic rehabilitated according to each case.

DETAILED DESCRIPTION:
Brånemark discovered the process of osseointegration in the 1960s and placed the first dental implant about 50 years ago. Since then dental implant became a basic alternative to conventional prosthodontic treatment options. Many clinical studies on dental implants have been published. Most studies present data on implant, prosthesis survival and on bone response adjacent to the implants. However, only few studies have investigated whether there is any possible correlation between serum levels of vitamin D and dental implant stability.

Osseointegration, the formation interface between implant and bone, is basic step of dental implant success. Although it depends on variety of causes mention some of them: surgical and prosthetic factors (surgical technique , operator experience, timing and type of prosthetic loading, and quality of prosthetic rehabilitation), implant-related factors (material, design, and surface), and patient-related factors (bone volume/quality at the recipient site and host response ). Mechanical stability of dental implant is a prerequisite for successful osseointegration. The alveolar bone architecture of the implant drilling site dictates the success of anchored endosseous dental implants. Immediately and up to several months afterwards, a series of cellular and molecular events occur where host tissues biologically integrate the alloplastic material into the native bony structure. As cortical bone withstand torsional loading and provides higher initial stability, cancellous bone is richer in vascular canals and thus, vasculature to supply mesenchymal progenitor cells. In this sense, the complex and dynamic process of osseointegration may occur via contact osteogenesis, where the implant surface is surrounded by bone cells after fixation to form de novo bone, or via distance osteogenesis, where bone formation is preceded by the osteoclastogenesis of the existing tissue. Despite all improvements introduced mainly on surgical and prosthetic protocols (design ,threads, micro- and nano-topographical (surface) treatments, and adding growth factors) all of them and more improve dental implant survival rate, making it possible to accomplish procedures were previously associated with high rate of failure as immediate implant placement and immediate load of dental implant. Meanwhile with such improvement but there are few percent of failure seem impossible to recognize its etiology. Based on chronological criteria, failures can be classified as either "early dental implant failures" (EDIFs) or "late dental implant failures" (LDIFs). EDIFs are due to unsuccessful osseointegration, indicating impaired bone healing, whereas LDIFs are due to loss of osseointegration. Both have different etiologies. LDIF is related to infection, occlusal overloading, and failure of the implant components. EDIF is usually caused by inadequate surgical and prosthetic protocols, low bone volume or quality at the recipient site, habits (smoking and parafunctions), or systemic conditions endanger osseointegration. Early failures due to lack of osseointegration are one of modern implantology nightmares. But as some patient categories seem to be specific vulnerable to it more than else, it might be possible to correlate it to patient's systemic health condition. Vitamin D is one of thi systemic condition that may have impact on dental implant failure but barely mentioned in dental literature. Today vitamin D is worldwide public health concern, vitamin D considered deficient when serum 25(OH) levels are <10 ng/mL, insufficient when serum levels are 10-30 ng/mL, and optimal with serum levels of >30 ng/mL. Vitamin D deficiency can result from inadequate dietary intake and insufficient exposure to sunlight. Vitamin D, fat-soluble hormone regulates calcium phosphate homeostasis and mineral bone metabolism. It is transformed into the active form (1, 25- dyhydroxy vitamin D3) by hydroxylation, firstly in the liver then in the kidney. It stimulates osteoblast bone matrix production, coupling bone resorption to form and optimize bone remodeling. As it increases calcium absorption in intestine and so reduce PTH secretion and systemic bone resorption with a possible inhibition of osteoclastogenesis. Vitamin D effect during dental implant osseointegration remains limited in literature. In animals, Kelly et al. studied the osseointegration process in rats with deficiency in Vitamin D and reported lower BIC values and mechanical bone strength after 2 weeks postimplant placement. Noteworthy that implant failure might be confounded by raise insufficiency of vitamin D prevalence in populations. Zhou et al. reported titanium screw fixation in rats after 8 weeks of oral treatment with vitamin D, with significant increment of peri-implant bone density, bone-implant contact (1.5 times higher) and peri-implant trabecular microarchitecture. Recently, topical application of vitamin D (10%) and melatonin (5%) solutions on the surface of immediate implants placed in dogs evaluated. Both topical applications significant improved new bone formation around implants and reduced crestal bone loss at 12 weeks following surgery, standing out positive correlation between vitamin D and early stages of osseointegration. Therefore, these results may suggest that vitamin D has effect on bone healing after implant insertion. Schulze-Spate et al., in a randomized, double-blind, placebo-controlled clinical trial in humans, reported finding a higher bone remodeling activity related to higher vitamin D levels. A retrospective study correlate early implant failure and low serum levels of vitamin D showed a higher incidence of the implant failure rate but a correlation between both factors could not determine . Therefore, vitamin D seems to improve bone health and implant healing. The present study will be selected from those seeking delayed dental implant selected from those attending the outpatient clinic at Oral and Maxillofacial Surgery Department in the Faculty of Dentistry, Ain Shams University from February 2020 to February 2021. The following data will be collected from each patient through diagnostic chart as follow: Personal data, chief complaint, full medical history, dental history, family history and personal habits as smoking, alcohol consumption and habits related to the oral hygiene. The study protocol will be explained to all prospective candidates, and a written informed consent will be received from each patient before participation. All the data will be reviewed by ethics commits of faculty of dentistry Ain Shams University.

Eligibility criteria:

I. Inclusion criteria:

1. Patients with vitamin D sufficient, insufficient and deficient according to Enzyme Immunoassay test.
2. Patients with horizontal ridge width and vertical ridge height, according to class III of Cawood and Howell classification.
3. Patients with matched parameters of implant including diameter, length and manufacturing.
4. Patients' compliance to oral hygiene measures.
5. Compliance with all requirements in the study and signing the informed consent.
6. Patient with sufficient inter arch space.

II. Exclusion criteria:

1. Patients with diseases of the immune system or any medical condition that may influence the outcome.
2. Patients with history of intravenous and/or oral bisphosphonate use.
3. Pathologic lesions in the site of implant placement.
4. Patients who are pregnant or lactating mothers.
5. Smokers patients.
6. Patients with poor oral hygiene habits that are not amenable to motivation and improvement.
7. Patients with history of irradiation of the head and neck region.
8. Patients who need pre-surgical augmentation for the alveolar ridge or sinus lift.
9. Patients need immediate implant placement. A-Pre-operative Phase 1- Clinical examination:

   * Clinical examination of the implant placement site for ensuring the health and amount of soft tissue.
   * Study models will have prepared and articulated to assess inter-arch space and analyze the occlusion with respect to the site of the future implant. 2- Radiographic examination:
   * Cone Beam Computed Tomography (CBCT) will be done for each patient to evaluate the alveolar ridge height and width at the site of implant placement. 3- Laboratory investigation: 25-hydroxy vitamin D level will be done for each patient preoperative using Enzyme Immunoassay (EIA) test categorized by mean serum vitamin D status as follows: [26]

     1. Sufficient, 25 (OH) D >30 ng/mL (>75 nmol/L)
     2. Insufficient, 25 (OH) D 10-30 ng/mL (50-75 nmol/L)
     3. Deficient, 25 (OH) D <10 ng/mL (<50 nmol/L). B- Surgical Phase
   * All patients will receive dental implants under local anesthesia according to the manufacturer drilling protocol.
   * The initial implant stability will be analyzed using Osstell® in terms of ISQ (Implant Stability Quotient) reading (R0). C-Post-operative Phase 1- Post-operative instructions:

Will be given for each patient in a written manner as follow:

* To apply ice packs, wrapped in a cloth to avoid frostbite, on the surgical site extra-orally for the first 24 hours (10 minutes every 30 minutes) to decrease edema.
* Following the first day, gentle rinsing by warm saline 3-5 times/day, for 1 week.
* To avoid vigorous gargling for the first 24 hours.
* To avoid hot food or drink for the first 24 hours. 2- Post-operative medications: Amoxicillin/Clavulanic acid 875mg/125mg oral tablet (Augmantin®) will prescribed twice daily for 5 days postoperatively (or Clindamycin 300 mg <Clindam®> in patients allergic to penicillin 3 times daily). [ Diclofenac potassium 50mg oral tablet (Cataflam®) three times daily for 3 days, and then whenever it's needed for pain relief and anti-inflammatory effect.
* Oral rinses with 0.125% Chlorohexidine HCL (Hexitol®) three times daily starting from the second day postoperatively and continued for two successive weeks. 3- Post-operative assessment:
* All patients will be recalled one week postoperatively to assess the overall healing process and ensure good oral hygiene. The sutures will be removed at this appointment.
* 12 weeks postoperatively (R12), all patients will be recalled to reassess the implant stability using Osstell® in terms of ISQ reading and each patient will receive the healing abutment after an adequate healing period according to the site of the implant in preparation for the prosthetic restoration.
* All patients will receive needed prosthetic restoration according to planned treatment plane. All data will be tabulated for statistical analysis to correlate Vitamin D serum level and ISQ readings (R0 and R12)

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with vitamin D sufficient, insufficient, and deficient according to Enzyme Immunoassay test. 2. Patients with horizontal ridge width and vertical ridge height, according to class III of Cawood and Howell classification. 3. Patients with matched parameters of implant including diameter, length and manufacturing. 4. Patients' compliance to oral hygiene measures. 5. Compliance with all requirements in the study and signing the informed consent. 6. Patient with sufficient inter arch space.

Exclusion Criteria:

* 1. Patients with diseases of the immune system or any medical condition that may influence the outcome. 2. Patients with history of intravenous and/or oral bisphosphonate use. 3. Pathologic lesions in the site of implant placement. 4. Patients who are pregnant or lactating mothers. 5. Smokers patients. 6. Patients with poor oral hygiene habits that are not amenable to motivation and improvement. 7. Patients with history of irradiation of the head and neck region. 8. Patients who need pre-surgical augmentation for the alveolar ridge or sinus lift. 9. Patients need immediate implant placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The present study will be selected from those seeking delayed dental implant selected from those attending the outpatient clinic at Oral and Maxillofacial Surgery Department in the Faculty of Dentistry, Ain Shams University from February 2020 to February 2021. The following data will be collected from each patient through diagnostic chart as follow: Personal data, chief complaint, full medical history, dental history, family history and personal habits as smoking, alcohol consumption and habits related to the oral hygiene. The study protocol will be explained to all prospective candidates, and a written informed consent will be received from each patient before participation. All the data will be reviewed by ethics commits of faculty of dentistry Ain Shams University.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2023-04-29 (Actual); Study Completion 2023-04-29 (Actual)

PRIMARY OUTCOMES:
early implant failure relation to vitamin D serum level | 12 weeks
  evaluation early implant failure within 3 months of implant placement using clinical and radiographic methods. implant consider failed if failed to osseointegrate without infection signs or failed with infection present showing signs of infection as pain, mobility, swelling and marginal bone loss more than 2.5 mm after 12 weeks of implant placement. Side by side with measuring implant stability at implant placement time and 12 weeks Laters. data were correlated with vitamin D serum levels.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Abd El-Raouf, BDS, Principal Investigator — Ain Shams University, Faculty of Dentistry
Locations (1):
- Faculty of dentistry Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided